CLINICAL TRIAL: NCT00003814
Title: Phase III Randomized, Double-Blind Study of DFMO vs. Placebo in Low Grade Superficial Bladder Cancer
Brief Title: Eflornithine in Treating Patients With Bladder Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000066966; ILEX-DFMO341; UCLA-9812049; UF-453-1998; WCCC-CO-98803; NCI-G99-1509
Record Dates: First submitted 1999-11-01; First posted 2004-02-20 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2007-05

CONDITIONS: Bladder Cancer
Keywords: stage 0 bladder cancer; stage I bladder cancer; recurrent bladder cancer; transitional cell carcinoma of the bladder
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Eflornithine

INTERVENTIONS:
Drug: eflornithine

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. It is not yet known if eflornithine is more effective than no further therapy in treating bladder cancer.

PURPOSE: Randomized phase III trial to determine the effectiveness of eflornithine in treating patients who have newly diagnosed or recurrent bladder cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine whether treatment with eflornithine is effective in preventing recurrence of tumor after transurethral resection in patients with low grade, superficial transitional cell carcinoma of the bladder. II. Determine the incidence and severity of toxicities associated with the long-term use of this drug in this patient population.

OUTLINE: This is a randomized, double blind, multicenter study. Patients are stratified according to disease status (newly diagnosed vs recurrent), clinical stage (Ta vs T1), grade (G1 vs G2), and focus (multifocal vs unifocal). Patients receive either oral eflornithine or placebo once daily. Treatment continues for 1 year in the absence of disease progression or unacceptable toxicity. Patients are followed every 3 months during the first 2 years, every 6 months for the third year, and then annually for the fourth year.

PROJECTED ACCRUAL: A total of 450 patients (225 per arm) will be accrued to this study within 1.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed low grade (grade 1 or 2), superficial (stage Ta or T1) transitional cell carcinoma (TCC) of the bladder Newly diagnosed or recurrent All visible tumor must have been resected within the past 12 weeks Standard clinical management determined to be expectant observation without further surgery, intravesical therapy, or systemic therapy No prior upper tract TCC No history of grade 3 TCC, carcinoma in situ including severe dysplasia, non-TCC histology, or TCC greater than or equal to T2 No involvement of upper urinary tract prior to or at the time of initial tumor resection Abdominal CT scan, IVP, or retrograde pyelogram within the past 3 months to rule out upper urinary tract tumor

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Not specified Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception No prior malignancy within the past 5 years and no concurrent malignancy except nonmelanomatous skin cancer or carcinoma in situ of the cervix No clinically significant hearing loss (i.e., hearing loss effects everyday life and/or wears a hearing aide) No other significant medical or psychiatric condition

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 4 weeks since prior growth factors No concurrent growth factors Chemotherapy: No prior systemic chemotherapy for bladder cancer No concurrent intravesical therapy At least 4 weeks since prior chemotherapy No concurrent chemotherapy Endocrine therapy: At least 4 weeks since prior high dose steroids or prednisone No concurrent high dose steroids No concurrent prednisone or its equivalent in excess of 10 mg/day Radiotherapy: No prior radiotherapy for bladder cancer At least 4 weeks since prior radiotherapy No concurrent radiotherapy Surgery: See Disease Characteristics Other: At least 4 weeks since prior carbamazepine or experimental drugs No concurrent carbamazepine or experimental drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 1999-02; Study Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Mayle, Study Chair — Genzyme, a Sanofi Company
Locations (61):
- United States (61):
  - Urology Associates, Birmingham, Alabama
  - Intouch Research, Huntsville, Alabama
  - Advanced Urology Medical Center, Anaheim, California
  - Citrus Valley Urological Medical Group, Glendora, California
  - University of California San Diego Cancer Center, La Jolla, California
  - San Diego Urology Center, La Mesa, California
  - South Coast Urological Medical Group, Laguna Hills, California
  - Foothill Urology Associates, Pasadena, California
  - San Bernadino Urological Associates, San Bernadino, California
  - DRC and Urological Physicians of San Diego, San Diego, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - Urology Specialists, P.C., Waterbury, Connecticut
  - George Washington University Hospital, Washington D.C., District of Columbia
  - Tampa Bay Meical Research, Clearwater, Florida
  - University of Florida - Gainesville, Gainesville, Florida
  - Urology Health Center, New Port Richey, Florida
  - Barzell, Whitmore, Treiman and Dunne - The Urology Treatment Center, Sarasota, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Piedmont Urology PC, Atlanta, Georgia
  - Georgia Urology, Atlanta, Georgia
  - Urology Associates, Inc., Marietta, Georgia
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - Wichita Clinic, P.A., Wichita, Kansas
  - 206 Research Associates, Greenbelt, Maryland
  - Mid Atlantic Clinical Research, Rockville, Maryland
  - Lahey Clinic - Burlington, Burlington, Massachusetts
  - Fallon Clinic, Inc., Worcester, Massachusetts
  - Urology Surgical Associates, Springfield, Missouri
  - Washington University Barnard Cancer Center, St Louis, Missouri
  - Office of Sheldon Freedman, Las Vegas, Nevada
  - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - University Hospital of New Mexico, Albuquerque, New Mexico
  - St. Joseph West Mesa Center, Albuquerque, New Mexico
  - Cancer Center of Albany Medical Center, Albany, New York
  - Veterans Affairs Medical Center - Albany, Albany, New York
  - Medical & Clinical Research Associates, LLC, Bay Shore, New York
  - Mount Sinai Medical Center, NY, New York, New York
  - University of Rochester Cancer Center, Rochester, New York
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - University of Oklahoma College of Medicine, Oklahoma City, Oklahoma
  - Oregon Cancer Center, Portland, Oregon
  - Earle A. Chiles Research Institute at Providence Portland Medical Center, Portland, Oregon
  - Kimmel Cancer Center of Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Allegheny University of the Health Sciences, Philadelphia, Pennsylvania
  - Albert Einstein Cancer Center, Philadelphia, Pennsylvania
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Urology Clinics of North Texas, Dallas, Texas
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - University of North Texas HSC, Fort Worth, Texas
  - Urology San Antonio Research, San Antonio, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Virginia Urology Center, Richmond, Virginia
  - Seattle Urological Associates, Seattle, Washington
  - Urology Northwest PS, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin